CLINICAL TRIAL: NCT05953259
Title: Randomised Controlled Clinical Trial to Evaluate STERN FIX Device as a Sternal Stabilization System in Patients After Sternotomy
Brief Title: RCT to Evaluate STERN FIX Device as a Sternal Stabilization System in Patients After Sternotomy
Acronym: FIXTER-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NEOS Surgery (Industry)
Collaborators: Hospital Clinic of Barcelona (Other); Complejo Hospitalario de Navarra (Other); Universitätsklinikum Freiburg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEO-SC1-2023-01
Record Dates: First submitted 2023-07-03; First posted 2023-07-20 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Median Sternotomy
Keywords: sternal closure; cardiac surgery; sternotomy
MeSH Terms: interventions — Bone Wires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and primary outcome assessors will not know whether the allocated sternotomy closure system is STERN FIX or wires only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STERN FIX (Active Comparator): Combination of at least one STERN FIX device and surgical wires to close median sternotomy (total of 5 fixation points)
  Interventions: Device: Combination of STERN FIX and wires
- Wires (Active Comparator): Standard of care median sternotomy closure method with surgical wires
  Interventions: Device: Wires

INTERVENTIONS:
Device: Combination of STERN FIX and wires — Closure of the median sternotomy using a combination of at least one STERN FIX device and wires for a total of 5 fixation points.
  Arms: STERN FIX
Device: Wires — Closure of the median sternotomy using the standard of care with steel wires.
  Arms: Wires

SUMMARY:
The goal of this clinical trial is to compare the safety and performance of the sternal stabilization system STERN FIX with the standard of care (sternal closure with wires only) in normal conditions of use, in patients of risk undergoing median sternotomy during cardiothoracic surgery. The main question it aims to answer is:

• whether STERN FIX is a safe and efficient device to close the sternum after a sternotomy in patients of risk, achieving higher sternal stability than wires one month after surgery Participants will have their median sternotomy closed using STERN FIX in combination with wires or wires only at the end of their cardiothoracic surgery, according to the allocated treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing surgery that requires median sternotomy
* Patients with at least one of the following risk criteria: obesity (BMI>30), diabetes, COPD, non serious osteoporosis (not associated with fractures), creatinine > 200 µmol/L and/or under dialysis treatment, scheduled Bilateral Internal Mammary Artery (BIMA) grafting
* Patients willing and capable of granting informed consent to participate in clinical research and who have granted written consent
* Patient willing and capable of complying with the protocol requirements

Exclusion Criteria:

* Patient with suspected or known allergies or intolerance to the device material (PEEK - polyether-ether-ketone and carbon fibre)
* Patient with insufficient quality or quantity of bone or any other serious structural bone damage at the sternum
* Patient with serious osteoporosis (associated with fractures) or a degenerative bone disease affecting the sternum
* Patients with a latent or active infection or inflammation at the surgical area, that according to the surgeon criteria may interfere in the device implantation or proper function.
* Patient with sternal anomalies that, according to the surgeon criteria, prevent the use of the product, such as bone tumours in the implantation area.
* Pregnant patients or patients planning to become pregnant during the first 6 months after surgery.
* Patients with diagnosis of dementia with a mental status score (MMSE) < 20.
* Patients with life expectancy lower than 6 months.
* Patients involved in other interventionist clinical trials or that have been involved in other interventionist clinical trials during the previous 4 weeks
* Parasternal sternotomy.
* Patients with intraoperative conditions that, according to the surgeon's opinion, require or exclude the use of a specific sternal closure system, or that cannot be closed following the study products instructions for use.

IMPORTANT: When the allocated closure method is wires only, the surgeon must assess whether the patient could have also had STERN FIX implanted in order to decide if the patient can continue in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sternal stability | 1 month after surgery
  The primary outcome of this study will evaluate the sternal stability through clinical assessment using the sternal instability scale (SIS) with grades 0 to 3 where 0 is "Clinically stable sternum" and 3 is "Completely separated sternum - entire length"

SECONDARY OUTCOMES:
Safety SAE/AE prevalence | 6 months after surgery
  All adverse events occurring during the study period will be recorded, except for frequent events after surgical interventions requiring median sternotomy.
Safety SAE/AE causality | 6 months after surgery
  All adverse events occurring during the study period will be recorded, except for frequent events after surgical interventions requiring median sternotomy.
Prevalence of device deficiencies | 6 months after surgery
  Adverse event related to the use of an investigational medical device. This includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction and events resulting from use error or from intentional misuse of the investigational medical device.
Reinterventions - prevalence | 6 months after surgery
  Prevalence of reinterventions
Reinterventions - Causality | 6 months after surgery
  Causality of reinterventions
Prevalence of sternal wound infections | 1 month and 6 months after surgery
  Prevalence of sternal superficial and deep wound infections
Prevalence of dehiscence | 1 month and 6 months after surgery
  Prevalence of dehiscence (without infection)
Sternal closure time | Surgery
  Measured time from the implantation of the first wire to the closure of the last wire (minutes)
Easiness of use of the closure method | Surgery
  The surgeon perceived difficulty of the sternal closure method will be recorded using the Likert scale (1 to 5).
Surgeon satisfaction of the closure method | Surgery
  General surgeon satisfaction with the sternotomy closure method will be recorded using the Likert scale (1 to 5).
Chest pain | Before surgery, 3 and 7 days postoperatively, during the first month and during 6 months postoperatively
  Patients will assess their chest pain using the NRS (0 to 10) while resting and after forced cough
Blood loss | During the first 12 hours postoperatively
  Total blood loss volume obtained from thoracic drainage during the first 12 hours postoperatively will be recorded (mL).
Upper Limb functional index | Before surgery, one month and 6 months postoperatively
  Patients will assess their upper limbs functional capacity using the Upper Limb functional index (ULFI-Sp)
Quality of life - EQ5D5L | Before surgery, one month and 6 months postoperatively
  Patients will complete the EQ-5D-5L questionnaire
Sternal halves union/malunion | 6 months after surgery
  Using CT scan images, the separation between the two sternal halves will be measured in mm. Later on, these measurements will be classified as:
  * Malunion: more than 3mm of separation
  * Mild malunion: between 1 and 3mm of separation
  * Union: less than 1mm of separation
Sternal halves alignment | 6 months after surgery
  Using CT scan images, the alignment between the two sternal halves will be assessed and classified as:
  * Misalignment: <50% alignment between sternal halves
  * Aligned: >50% de alignment between halves
Sternum integrity | 6 months after surgery
  Using CT scan images, the presence of bone cuts, fractures or necrosis will be assessed.
Closure system integrity | 6 months after surgery
  Using CT scan images, the sternal closure devices integrity will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Manel Castellà Pericás, MD/PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (5):
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Spain (4):
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville